CLINICAL TRIAL: NCT04364945
Title: Association Between Anesthetic Drugs for General Anesthesia and Postoperative Intelligence/behavioral Assessment Results in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H2003-234-1115
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia and Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Dexmedetomidine; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): General anesthesia is maintained using sevoflurane only. Sevoflurane concentration is adjusted to maintain bispectral index value between 40 and 60.
  Interventions: Drug: Sevoflurane
- Dexmedetomidine-remifentanil(DEX-R) group (Experimental): General anesthesia is maintained using sevoflurane, dexmedetomidine (1 mcg/kg loading, and 1 mcg/kg/hr continuous infusion) and remifentanil (0.1-0.2 mcg/kg/min). Sevoflurane concentration is adjusted to maintain bispectral index value between 40 and 60.
  Interventions: Drug: dexmedetomidine; Drug: remifentanil; Drug: Sevoflurane

INTERVENTIONS:
Drug: dexmedetomidine — administration of dexmedetomidine 1 mcg/kg/hr
  Arms: Dexmedetomidine-remifentanil(DEX-R) group
Drug: remifentanil — administration of remifentanil 0.1-0.2 mcg/kg/min
  Arms: Dexmedetomidine-remifentanil(DEX-R) group
Drug: Sevoflurane — Anesthesia is maintained using sevoflurane.

SUMMARY:
In this study, we compared the results of the intelligence and behavioral test performed after surgery between the group using sevoflurane and the group receiving dexmedetomidine and remifentanil, in Korean children under 2 years of age who underwent surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children under 2 years of age who underwent general anesthesia for elective surgeries inlcuding urology, surgery, plastic surgery, orthopedics, and otolaryngology, etc, which were non-staged and non-repetitive procedures
* American Society of Anesthesiology Physical Status I, II

Exclusion Criteria:

* Allergies to narcotic analgesics
* With massive bleeding or shock
* Heart, lung, kidney or liver disease
* Central / peripheral nervous system disease and disorder
* Any physical deformity and disorder, genetic disease, chromosomal disease
* Previous history of general anesthesia or sedation
* Developmental delay identified through K-DST results
* Additional exposure to general anesthetics or sedative drugs during follow-up

Ages: 1 Month to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Wechsler Preschool and Primary Scale of Intelligence-IV at age of 5 | When the patient's age is 5 years after surgery
  categorization: 130 and above: Very Superior 120-129: Superior 110-119: High Average 90-109: Average 80-89: Low Average 70-79: Borderline

SECONDARY OUTCOMES:
Leiter International Performance Scale at age of 30 months | When the patient's age is 30 months old after surgery
  Korean version of the Leiter International Performance Scale-Revised (Leiter-R), categorization:
  130 and above: Very Superior 120-129: Superior 110-119: High Average 90-109: Average 80-89: Low Average 70-79: Borderline
Wechsler Preschool and Primary Scale of Intelligence-IV at age of 7 | When the patient's age is 7 years old after surgery
  categorization: 130 and above: Very Superior 120-129: Superior 110-119: High Average 90-109: Average 80-89: Low Average 70-79: Borderline
Child Behavior Checklist results | When the patient's age become 30 months, 5 years and 7 years old after surgery
  Child Behavior Checklist results at age of 30 months, 5 years and 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hyun Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Other, South Korea

REFERENCES:
- [Derived] Ji SH, Kang P, Cho SA, Park JB, Jang YE, Kim EH, Kim JT, Kim HS, Jung HJ, Jung HA, Lee HC, Lee JH. Effects of Dexmedetomidine-Remifentanil on Neurodevelopment of Children after Inhalation Anesthesia: A Randomized Clinical Trial. Anesthesiology. 2025 Oct 1;143(4):827-834. doi: 10.1097/ALN.0000000000005634. Epub 2025 Sep 9. PMID 40923823